CLINICAL TRIAL: NCT06628895
Title: Effect of Modified Poco-Poco Exercise to Frailty Stages, Expression of Global DNA Methylation, GDF15 and Lamin A COP on Elderly Living On Community in Bandung
Brief Title: Effect of Modified Poco-Poco Exercise to Frailty Stages, Expression of Global DNA Methylation, GDF15 and Lamin A COP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IKFR-202410.01
Record Dates: First submitted 2024-09-26; First posted 2024-10-08 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Frail Elderly
MeSH Terms: interventions — Exercise; Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Frail elderly living in community (Experimental): Adult above 60 years old, frailty level based on Fried frailty phenotype, without having diabetes mellitus and cardiac disease
  Interventions: Other: EXERCISE TRAINING WITH OR WITHOUT MEDICATION

INTERVENTIONS:
Other: EXERCISE TRAINING WITH OR WITHOUT MEDICATION — Exercise training that consists of flexibility, aerobic, balance and strengthening regime. The exercise given three times a week, for 12 weeks.

SUMMARY:
The goal of this clinical trial is to know the effect of multicomponent exercise in frail elderly in community to aging hallmarks. The main question[s] it aims to answer are:

1. Do global DNA methylation levels change in elderly people in Bandung after receiving modified poco-poco exercise?
2. Do GDF15 levels change in elderly people in Bandung after they are given modified poco-poco exercise?
3. Do lamin A COP levels change in elderly people in Bandung after they are given modified poco-poco exercise?
4. Does the level of frailty in elderly people in Bandung change after they are given modified poco-poco exercise?

Participants will be asked to do flexibility, balance, aerobic and strengthening exercise included in poco-poco modified exercise three times a week for 12 weeks

DETAILED DESCRIPTION:
The elderly population in West Java Province with the age category of 60-64 years is 1.76 million people. Experts estimate that 25.2% of the Indonesian population experiences frailty. Frailty can lead to a variety of worsening health conditions. The frailty process is thought to stem from the failure of various mechanisms associated with markers of aging. Markers of aging are divided into three categories: primary, antagonistic and integrative. Biomarkers representing these three categories are global DNA methylation, GDF15 and Lamin A COP. Multicomponent exercise is the most effective intervention in elderly with frailty. Elderly people in West Java on average only have an education equivalent to junior high school (SMP), so activities that promote physical activity are better focused on health activities in the community. The poco-poco exercise that is currently commonly practiced almost fulfills the rules of multicomponent exercise for frailty elderly, but poco-poco exercise does not have a muscle strengthening exercise component, so a modified poco-pcoco exercise was created to fulfill this method.

ELIGIBILITY:
Inclusion Criteria:

1. Frailty level is in pre-frailty
2. MoCA INA score above 18
3. Domicile in Bandung City
4. Willing to participate in the study after informed consent

Exclusion Criteria:

1. There is a hearing impairment that may prevent the subject from receiving verbal instructions
2. There is uncorrected visual impairment
3. There are musculoskeletal disorders so that they cannot perform exercise procedures or procedures for measuring research variables
4. Subjects received other rehabilitation programs
5. Post-stroke with average limb muscle strength below three
6. There are diseases that cause impaired cognition such as Alzheimer's disease, traumatic head injury, Parkinson's disease.
7. There are severe joint diseases such as osteoarthritis and rheumatoid arthritis that may worsen during exercise or may cause difficulty in carrying out the exercise program.
8. Severe cardiovascular disease as assessed by a heart and vascular specialist
9. Unable to attend Exercises regularly

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Level of Global DNA Methylation in 12 Weeks | week 0 and week 12
  Global DNA Methylation will be measured twice using ...
Change From Baseline in Level of Growth Deficiency Factor (GDF15) in 12 Weeks | week 0 and week 12
  GDF15 will be measured using blood plasma with Enzyme Linked Immuno Assay (ELISA), expected GDF value that show improvement that it will be decreased
Change From Baseline in Level of Lamin A (Cyclic Osteo Progenitor) COP in 12 Weeks | week 0 and week 12
  Lamin A COP will be measured with flow cytometry from Peripheral Blood Mononuclear Cells (PBMC), the value that shows improvement has a lesser lamin A COP population
Change From Baseline in Level of Frailty in 12 Weeks | week 0 and week 12
  Level of Frailty is measured using Fried's Frailty Phenotype with range 1-5 with 5 is the worst level of frailty. Fried's frailty measured with five components that are unintentional weight loss, muscle weakness, exhaustion on activity, slow gait and low physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Irma R. Defi, DR. Med. Sc, dr, SpKFR, Ger(K), Study Director — Faculty of Medicine Universitas Padjadjaran
Locations (1):
- Puskesmas Sekejati, Bandung, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No